CLINICAL TRIAL: NCT07281924
Title: A Phase 1b/2 Trial Evaluating the Safety, Tolerability, and Preliminary Efficacy of Melphalan Percutaneous Hepatic Perfusion Therapy (HEPZATO KIT™) With Nivolumab and Relatlimab (Opdualag) in Patients With Metastatic Melanoma and Liver Metastasis
Brief Title: Hepzato Kit and Opdualag for Metastatic Melanoma and Liver Metastasis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1424; UW25072 (Other: OnCore ID); Protocol Version 9/26/25 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Melanoma; Liver Metastases
Keywords: immunotherapy; Liver metastases; Anti-PD-1; Anti-LAG-3; Melphalan; Percutaneous Hepatic Perfusion Therapy; Liver directed therapy; Nivolumab; Relatlimab; Immune Checkpoint Inhibitors; Hepzato; Opdualag
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; relatlimab; Opdualag

STUDY DESIGN:
Intervention Model Description: Five patients will be treated first. If at least two achieve an objective response and no more than two experience a DLT, an additional ten patients will be enrolled, giving a total sample of fifteen. If the first 5 participants records three or more DLTs, or one or fewer responses, the trial will halt.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Metastatic Melanoma (Experimental)
  Interventions: Drug: Nivolumab and Relatlimab; Device: Melphalan

INTERVENTIONS:
Drug: Nivolumab and Relatlimab — Relatlimab is a human IgG4 LAG-3 blocking antibody. Nivolumab is a human IgG4 PD-1 blocking antibody. Nivolumab 480 mg and relatlimab 160 mg in a fixed-dose combination will be administered on Day 1 of each 28-day cycle that the participant is on treatment and will be given for up to 2 years from start of treatment.
  Other Names: Opdualag
Device: Melphalan — The recommended HEPZATO dose is 3 mg/kg based on ideal body weight (IBW), infusion every 6 to 8 weeks for up to 2 total infusions
  Other Names: HEPZATO KIT

SUMMARY:
This study is being done to see if combining HEPZATO KIT™ with nivolumab and relatlimab (Opdualag™) in the first line setting in patients with metastatic melanoma with liver metastasis is safe, tolerable, and will have a synergistic effect leading to improved clinical outcomes compared to the historic cohort of patients with liver metastasis treated with combination immune checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
Co-Primary Objectives

* To evaluate the safety and tolerability of HEPZATO KIT™ in combination with nivolumab and relatlimab (Opdualag™) in subjects with metastatic melanoma and liver metastasis (LM).
* To evaluate the preliminary systemic efficacy of HEPZATO KIT™ in combination with nivolumab and relatlimab (Opdualag™), as measured by objective response rate (ORR), in subjects with metastatic melanoma and LM.

Secondary Objectives

* To evaluate the preliminary systemic efficacy of HEPZATO KIT™ in combination with nivolumab and relatlimab (Opdualag™), as measured by ORR, in both hepatic and non-hepatic target lesions in subjects with metastatic melanoma and LM.
* To evaluate the disease control rate (DCR) in subjects with metastatic melanoma and LM receiving HEPZATO KIT™ in combination with nivolumab and relatlimab (Opdualag™).
* To evaluate the PFS in subjects with metastatic melanoma and LM receiving HEPZATO KIT™ in combination with nivolumab and relatlimab (Opdualag™).
* To evaluate the overall survival (OS) in subjects with metastatic melanoma and LM receiving HEPZATO KIT™ in combination with nivolumab and relatlimab (Opdualag™).
* To evaluate the duration of response (DOR) in subjects with metastatic melanoma and LM receiving HEPZATO KIT™ in combination with nivolumab and relatlimab (Opdualag™).
* To evaluate the tumor reduction at any time during treatment in subjects with metastatic melanoma and LM receiving HEPZATO KIT™ in combination with nivolumab and relatlimab (Opdualag™).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic melanoma with liver metastasis (LM). Liver biopsy positive for presence of melanoma metastases is required.
* Systemic treatment naïve in the unresectable/metastatic setting - prior adjuvant anti-programmed cell death-1 (anti-PD-1) and BRAF/MEK targeted therapy is allowed but must be greater than 6 months from the last treatment.
* Evaluable/measurable disease according to RECIST v1.1.
* Demonstrate adequate organ function; all screening labs to be obtained within 28 days prior to registration.
* Patients must weigh greater than or equal to 35 kilograms (due to possible size limitations with respect to percutaneous catheterization of the femoral artery and vein using the Delcath Hepatic Delivery System).

Exclusion Criteria:

* Prior treatment with HEPZATO KIT™ or nivolumab and relatlimab (Opdualag™)
* Radiotherapy is permitted within 30 days prior to C1D1 as long as radiation is given with palliative intent and towards a non-target lesion.
* History of hypersensitivity or treatment discontinuation due to grade 3+ immune-related adverse events (irAEs) from prior anti-PD-(L)1 therapy. Patients who are able to successfully resume immune checkpoint therapy without recurrence of grade 3 irAEs are eligible to participate.
* Symptomatic or uncontrolled brain metastases, leptomeningeal disease, or spinal cord compression not definitively treated with surgery or radiation.
* Prednisone use greater than or equal to 10 mg/d or equivalent
* Organ transplant recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Dose Limiting Toxicities (DLTs) | up to 12 weeks
  A DLT is defined as any grade 4+ non-hematologic event lasting greater than 3 days (despite appropriate medical management) considered possibly related to study treatment (HEPZATO KIT™ or Opdualag™) within 12 weeks of Cycle 1 Day 1.
Incidence of Treatment-Emergent Adverse Events | up to 2 years
Incidence of Serious Treatment-Emergent Adverse Events | up to 2 years
Number of Participants that Discontinue Treatment due to Adverse Events | up to 2 years
Overall Response Rate (ORR) | After treatment plus follow up for 2 years (up to 4 years)
  The objective response rate is the proportion of all participants with confirmed Partial Response (PR) or Complete Response (CR) according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).

SECONDARY OUTCOMES:
ORR in Hepatic and Non-Hepatic Lesions | After treatment plus follow up for 2 years (up to 4 years)
  The proportion of all participants with confirmed PR or CR according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment) in Hepatic and Non-Hepatic Target Lesions.
Disease Control Rate (DCR) | After treatment plus follow up for 2 years (up to 4 years)
  The disease control rate is the proportion of all subjects with SD for 8 weeks, or PR, or CR according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).
Progression Free Survival (PFS) | After treatment plus follow up for 2 years (up to 4 years)
  A measurement from the date of randomization until the criteria for disease progression is met as defined by RECIST 1.1 or death occurs. Participants who have not progressed will be right-censored at the date of the last disease evaluation.
Overall Survival (OS) | After treatment plus follow up for 2 years (up to 4 years)
  Overall survival is defined by the date of randomization to date of death from any cause.
Duration of Response (DOR) | After treatment plus follow up for 2 years (up to 4 years)
  Duration of overall response-the period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since treatment started).
Number of Participants with Tumor Reduction at any time | After treatment plus follow up for 2 years (up to 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ma, MD, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers must have local IRB approval for their study that is to include study of the biospecimens and accompanying data. Release of biospecimens to non-UW researchers will be performed according to all UW regulatory policies. Tissue (including blood) specimen as part of this research will be primarily stored at UW and may be sent to an outside lab/facility to achieve the objectives of the study. No study data or patient health information will be shared with a third party.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Researchers who are doing biomedical research may apply to the PI for access to blood and tissue (no patient identifiers on tubes or slides). Only de-identified information will be released with the specimens